CLINICAL TRIAL: NCT07211789
Title: Real World Evidence en Pacientes pediátricos Con Enfermedad de Crohn Activa
Brief Title: Real World Evidence Study With Restrictive Diet and Otral Nutritional Supplementation on Pediatric Patients With Active Chron Disease
Acronym: REVIDEC
Status: Completed | Type: Observational
Sponsor: Outcomes'10 (Network)
Collaborators: Nestlé Health Science Spain (Industry)
Responsible Party: Sponsor
Other Study IDs: NES-2019-050-OBS-CROHN
Record Dates: First submitted 2025-10-01; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Crohn Disease
Keywords: Inflammatory Bowel Disease; Pediatric Crohn's Disease; Children; Pediatrics; Observational Study; Multicenter Study; Prospective Study; Quality of Life; exclusion diet; wPCDAI; MINI index
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Pediatric Crohn's disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 8-18 years with Crohn's disease initiating treatment with EEN+CDED

SUMMARY:
This prospective study aims to provide real-world evidence of the effectiveness of the NEP + CDED diet in paediatric patients with Crohn's disease under conditions of routine clinical practice.

DETAILED DESCRIPTION:
Pediatric Crohn's disease is a chronic inflammatory disorder of the gastrointestinal tract that impacts growth and quality of life. Exclusive enteral nutrition (EEN) is the standard dietary treatment to induce remission, although its use is limited by low acceptability and strict dietary restrictions.

The combination of partial enteral nutrition (PEN) with the Crohn's Disease Exclusion Diet (CDED) represents a more tolerable alternative that reduces exposure to harmful dietary components and has shown efficacy in inducing clinical remission in previous studies.

This observational, prospective, multicenter study will evaluate the effectiveness of CDED+PEN in routine clinical practice in pediatric patients (8-18 years) with active Crohn's disease. The primary objective is to assess the proportion of patients achieving clinical remission (wPCDAI ≤ 12.5) and mucosal healing (MINI Index < 8), steroid-free at weeks 6, 12, and 24, and anti-TNF-free at week 24.

Secondary objectives include assessing health-related quality of life (IMPACT-III), treatment satisfaction and gastrointestinal tolerance, treatment persistence, and estimation of healthcare resource utilization and associated costs. The study is observational, descriptive, and non-interventional with respect to drugs, and will be conducted in pediatric patients initiating CDED+PEN as part of standard clinical care. Treatment prescription will be independent of study participation, and patients who receive the indication may be invited to participate after providing informed consent together with their parents or legal guardians.

Primary outcome measures include the frequency of patients in steroid-free clinical remission at weeks 6, 12, and 24, anti-TNF-free remission at week 24, and the proportion achieving mucosal healing (MINI Index < 8) at the same time points. Secondary analyses will include quality of life scores (IMPACT-III), distribution of questionnaire responses on satisfaction and tolerance, treatment persistence assessed by survival analysis, and cost estimates based on healthcare resource use.

This study will provide real-world evidence on the effectiveness, acceptability, and sustainability of the dietary approach with CDED+PEN in pediatric Crohn's disease under routine clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease (diagnosis based on clinical, laboratory, endoscopic, radiological, and histological criteria, according to the revised Porto criteria of the ESPGHAN for the diagnosis of inflammatory bowel disease in children and adolescents);
* Aged between 8 and 18 years;
* Who are about to start treatment with NEP + CDED, i.e. CDED-naive patients who may have previously received treatment with NEE;
* With active Crohn's disease defined by the Weighted Paediatric Crohn's Disease Activity Index (wPCDAI) ≥ 12.5;
* With data collection available for the following 6 months;
* Able to follow the study protocol or whose parent/caregiver is able to adhere to the study protocol, according to the investigator's perspective.

Exclusion Criteria:

* Patients with ulcerative colitis and/or unclassified inflammatory bowel disease.
* Patients with more than 36 months of disease progression.
* Penetrating (B3) and/or non-inflammatory stenosing (B2) pattern.
* Active perianal disease.
* Presence of extraintestinal manifestations.
* Patients who, in the investigator's opinion, will require surgical treatment or initiation of steroids or biological drugs (anti-TNF, vedolizumab or ustekinumab) within the next 3 months and for whom nutritional support is indicated exclusively as a bridge. Patients who are undergoing biological treatment but discontinue treatment due to non-response and initiate CDED+NEP are not excluded.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 8-18 years with Crohn's disease initiating treatment with exclusive enteral nutrition (EEN) plus the Crohn's Disease Exclusion Diet (CDED) and whose wPCDAI value is equal to or greater than 12.5.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the CDED + NEP | Weeks 6, 12, 24
  Measurement of absolute and relative frequencies of patients in steroid-free remission
Effectiveness of the CDED + NEP | At week 24
  Measurement of absolute and relative frequencies of patients in anti-TNF-free remission
Mucosal healing | Weeks 6, 12, 24
  The relative and absolute frequencies of patients who have obtained a score of <8 on the MINI Index will be calculated; this value implies healing of the mucosa.

SECONDARY OUTCOMES:
Health-related quality of life | Weeks 6, 12, 24
  The scores obtained with the HRQoL questionnaire will be calculated
Satisfaction and acceptability with nutritional treatment | Weeks 6, 12, 24
  Based on the distribution of responses to the questionnaire items
Gastrointestinal tolerance | Weeks 6, 12, 24
  Distribution of responses to questionnaire items
Persistence with the diet | Weeks 6, 12, 24
  Percentage of patients who persist with the diet at
Healthcare resource use and associated costs | Weeks 6, 12, 24
  It will be calculated:
  * Number of visits to professionals who treat the patient (specialist in gastroenterology and paediatric nutrition, primary care, nursing, educational psychologist, social worker, dietitian/nutritionist)
  * Number of visits to the emergency room per month,
  * Number of days hospitalised per month,
  * Number of complementary tests per month,
  * Number of days of sick leave taken by the caregiver per month,
  * Number of school days missed per month.
  For each patient, the monthly cost associated with the use of resources will be estimated by multiplying the frequency of use per month of each resource by its unit cost. Unit costs will be extracted from eSalud.

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital Torrecárdenas, Almería
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Univeristari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Materno-Infantil de Canarias de Las Palmas, Las Palmas de Gran Canaria
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Niño Jesús, Madrid
  - Hospital Universitario Materno Infantil, Málaga
  - Hospital Universitario Central, Oviedo
  - Hospital Universitario de Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario la Fe, Valencia

IPD SHARING:
Plan to Share IPD: No